CLINICAL TRIAL: NCT00839800
Title: A Comparison of Symbicort® SMART (160/4.5μg) and Symbicort® Turbuhaler 160/4.5 μg, Plus Terbutaline Turbuhaler 0.4 mg as Needed, for Treatment of Asthma - a 12-month, Randomized, Double-blind, Parallel Group, Active-controlled, Multinational Phase III Study in Asthmatic Patients From 16 Years
Brief Title: Study to Investigate the Efficacy of Symbicort® SMART.
Acronym: SAKURA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D589LC00001
Record Dates: First submitted 2009-02-04; First posted 2009-02-10 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: Asthma; Symbicort Turbuhaler
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Symbicort Turbuhaler 160/4.5 µg one inhalation bid (twice daily) + Symbicort Turbuhaler 160/4.5 µg as needed
  Interventions: Drug: Symbicort Turbuhaler
- 2 (Active Comparator): Symbicort Turbuhaler 160/4.5 µg one inhalation bid (twice daily) + terbutaline Turbuhaler 0.4 mg as needed
  Interventions: Drug: Symbicort Turbuhaler; Drug: Terbutaline Turbuhaler

INTERVENTIONS:
Drug: Symbicort Turbuhaler — 160/4.5 µg
Drug: Terbutaline Turbuhaler — 0.4 mg
  Arms: 2

SUMMARY:
The primary objective of this study is to compare the efficacy of Symbicort SMART (Symbicort Turbuhaler 160/4.5μg, one inhalation twice daily plus as needed) with Symbicort Turbuhaler 160/4.5μg, one inhalation twice daily plus terbutaline Turbuhaler 0.4 mg as needed, as asthma therapy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma according to the Global Initiative for Asthma guidelines (GINA) 2007 with a documented history of at least 6 months duration.
* Reversible airway obstruction, defined as an increase in FEV1 ≥12% relative to baseline for all patients 15-30 minutes after inhalation of in total 2 x 0.4 mg terbutaline Turbuhaler
* Prescribed use of inhaled glucocorticoid steroid (GCS) (any brand) for at least 12 weeks.

Exclusion Criteria:

* Respiratory infection affecting the asthma, as judged by the investigator, within 4 weeks.
* Intake of oral, rectal or parenteral GCS within 4 weeks and/or depot parenteral GCS within 12 weeks.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2091 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Andersson, MD, Study Director — AstraZeneca R&D Lund; Tito Atienza, M.D., Principal Investigator — Mary Mediatrix Medical Center, Lipa City, Philippines
Locations (109):
- Argentina (9):
  - Research Site, Buenos Aires, Argentina
  - Research Site, Capital Federal, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Monte Grande, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Santa Fe, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Ciudad de Buenos Aires
- Brazil (7):
  - Research Site, Porto Alegre, Brasil
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Juiz de Fora, Minas Gerais
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Florianópolis, Santa Catarina
  - Research Site, Santo André, São Paulo
- China (8):
  - Research Site, Shenyang, Liaoning
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Nanjing
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Xi'an
- Costa Rica (2):
  - Research Site, Tres Ríos, Cartago Province
  - Research Site, Barrio San Bosco, Provincia de San José
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Deszk
  - Research Site, Gyula
  - Research Site, Nyíregyháza
  - Research Site, Százhalombatta
- India (10):
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Mysore, Karnataka
  - Research Site, Trivandrum, Kerala
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Jaipur, Rajasthan
  - Research Site, Coimabatore, Tamil Nadu
  - Research Site, Noida
- Japan (45):
  - Research Site, Komaki, Aichi-ken
  - Research Site, Seto, Aichi-ken
  - Research Site, Asahi, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyushu, Fukuoka
  - Research Site, Yanagawa, Fukuoka
  - Research Site, Isesaki, Gunma
  - Research Site, Ōwa, Gunma
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Chitose, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tomakomai, Hokkaido
  - Research Site, Ako, Hyōgo
  - Research Site, Himeji, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Hitachi, Ibaraki
  - Research Site, Naka-gun, Ibaraki
  - Research Site, Morioka, Iwate
  - Research Site, Sakaidechō, Kagawa-ken
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Kawasaki, Kanagawa
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kochi, Kochi
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Nagaoka, Niigata
  - Research Site, Niigata, Niigata
  - Research Site, Beppu, Oita Prefecture
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Kurashiki, Okayama-ken
  - Research Site, Okayama, Okayama-ken
  - Research Site, Sakai, Osaka
  - Research Site, Matsue, Shimane
  - Research Site, Utsunomiya, Tochigi
  - Research Site, Chūō, Tokyo
  - Research Site, Kodaira, Tokyo
  - Research Site, Kokubunji, Tokyo
  - Research Site, Machida, Tokyo
  - Research Site, Nakano-ku, Tokyo
  - Research Site, tabashi City, Tokyo
  - Research Site, Toshima-ku, Tokyo
- Malaysia (5):
  - Research Site, Kubang Kerian, Kelantan
  - Research Site, Kuantan, Pahang
  - Research Site, Batu Caves, Selangor
  - Research Site, George Town
  - Research Site, Kuala Lumpur
- Peru (2):
  - Research Site, Lima, Lima Province
  - Research Site, Surco, Lima region
- Philippines (5):
  - Research Site, Lipa City, Batangas
  - Research Site, Davao City, Philippines
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Quezon City
- South Korea (4):
  - Research Site, Bucheon-si
  - Research Site, Cheongju-si
  - Research Site, Seoul
  - Research Site, Suwon
- Thailand (5):
  - Research Site, Bangkoknoi, Bangkok
  - Research Site, Hat Yai, Changwat Songkhla
  - Research Site, Naimuang, Nakhonratchasima
  - Research Site, Bangkok, Thailand
  - Research Site, Khon Kaen

REFERENCES:
- [Derived] Zhang O, Minku LL, Gonem S. Detecting asthma exacerbations using daily home monitoring and machine learning. J Asthma. 2021 Nov;58(11):1518-1527. doi: 10.1080/02770903.2020.1802746. Epub 2020 Aug 14. PMID 32718193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant entered the study on 16 February 2009, and the last participant completed the study on 23 February 2011. A total of 3209 participants were enrolled at 148 centres in 13 countries in Asia, America and Europe, and 2091 participants who fulfilled the randomisation criteria were randomised.
Pre-assignment Details: The study started with an enrolment visit, Visit 1, 1-7 days prior to Visit 2 (run-in). At Visit 2 patients had to have a reversibility of ≥12% relative to baseline and their pre-bronchodilatory Forced expiratory volume in one second (FEV1) had to be ≥50% of the predicted normal value.
Groups:
- Symbicort SMART: Symbicort Turbuhaler 160/4.5 microgram (mcg) one inhalation twice daily (bid) + Symbicort Turbuhaler 160/4.5 mcg as needed
- Symbicort+Terbutaline As Needed: Symbicort Turbuhaler 160/4.5 mcg one inhalation twice daily + terbutaline Turbuhaler 0.4 mg as needed
Period: Overall Study
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Started | 1049 | 1042
Completed | 956 | 932
Not Completed | 93 | 110
Not completed — Adverse Event | 8 | 12
Not completed — Lost to Follow-up | 31 | 26
Not completed — Withdrawal by Subject | 28 | 34
Not completed — Incorrect Enrolment | 3 | 3
Not completed — Study-Specific Discontinuation Criteria | 6 | 13
Not completed — Safety Reasons | 2 | 1
Not completed — Other | 8 | 14
Not completed — Severe Non-Compliance to Protocol | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed | Total
Number analyzed (Participants) | 1049 | 1042 | 2091
Age Continuous [Mean (Full Range); unit: years] | 45.7 [16 to 84] | 45.6 [16 to 85] | 45.7 [16 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 722 | 692 | 1414
  Male | 327 | 350 | 677

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Had Experienced Asthma Exacerbation(s) at the End of the Study
Description: Asthma exacerbation was defined as deterioration in asthma leading to oral glucocorticosteroid [GCS] treatment, hospitalization, or emergency room [ER] treatment.
Time Frame: week 52
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Number; unit: percentage of participants
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1049 | 1042
percentage of participants | 16 | 22

2. Secondary Outcome: Number of Asthma Exacerbations
Description: Asthma exacerbation was defined as deterioration in asthma leading to oral GCS treatment, hospitalization, or ER treatment. Number of asthma exacerbations during 52 weeks treatment was presented here.
Time Frame: up to 52 weeks
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Number; unit: Asthma exacerbations
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1049 | 1042
Asthma exacerbations | 259 | 363

3. Secondary Outcome: Morning Peak Expiratory Flow (PEF)
Description: The mean value from a 52-week treatment period.
Time Frame: 52-week treatment period
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Mean (Standard Deviation); unit: Liter/minute (L/min)
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1034 | 1026
Liter/minute (L/min) | 331.8 (102.2) | 324.7 (101.9)

4. Secondary Outcome: Evening PEF
Description: The mean value from a 52-week treatment period.
Time Frame: 2-week run-in period (14 - 18 days before randomization - week 0) and a 52-week treatment period
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1034 | 1026
L/min | 334.2 (102.6) | 327.8 (103.1)

5. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: The mean value for Weeks 4, 12, 24, 36 and 52 was analysed.
Time Frame: 4, 12, 24, 36 and 52 weeks after randomization
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Geometric Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1049 | 1042
Liter (L) | 2.258 (0.76) [NA to NA] | 2.222 (0.77) [NA to NA]

6. Secondary Outcome: Use of As-needed Medication
Description: The mean value of total daily number of inhalations from the treatment period for use of as-needed medication (daytime, night-time).
Time Frame: 52-week treatment period
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Mean (Standard Deviation); unit: inhalations/day
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1032 | 1026
inhalations/day | 1.21 (1.39) | 1.46 (1.60)

7. Secondary Outcome: Asthma Symptom Score
Description: The mean value from the treatment period for Total Asthma Symptom Score (total score: 0 is best - no asthma symptoms; 6 is worst).
Time Frame: 52-week treatment period
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1034 | 1025
units on a scale | 1.12 (1.04) | 1.22 (1.02)

8. Secondary Outcome: Nights With Awakening(s) Due to Asthma Symptoms
Description: The mean value from the treatment period was presented here.
Time Frame: 52-week treatment period
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Mean (Standard Deviation); unit: Nights With Awakening(s)
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1024 | 1025
Nights With Awakening(s) | 15.7 (27.1) | 17.5 (27.2)

9. Secondary Outcome: The Percentage of Participants Who Had Experienced First Mild Asthma Exacerbations
Description: Mild asthma exacerbation was defined as morning PEF ≥20% below baseline, daily as-needed medication use ≥2 inhalations above baseline, or a night with awakening due to asthma symptoms. The percentage of participants who had experienced mild asthma exacerbation(s) at the end of the study was presented here.
Time Frame: up to 52 weeks
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Number; unit: percentage of participants
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1049 | 1042
percentage of participants | 71 | 80

10. Secondary Outcome: Symptom-free Days (no Symptoms and no Awakenings)
Description: A symptom-free day was defined as a day without daytime or night-time symptoms and without night-time awakenings due to asthma symptoms. The mean value was presented here.
Time Frame: 52-week treatment period
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Mean (Standard Deviation); unit: symptom-free days
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1034 | 1026
symptom-free days | 45.5 (37.8) | 41.6 (37.2)

11. Secondary Outcome: Percentage of As-needed-free Days
Description: An as-needed-free day is defined as a night and day with no use of as-needed medication. The mean value from the treatment period was presented here.
Time Frame: 52-week treatment period
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Mean (Standard Deviation); unit: percentage of as-needed-free days
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1032 | 1026
percentage of as-needed-free days | 51.4 (36.7) | 47.2 (36.7)

12. Secondary Outcome: Percentage of Asthma-control Days (no Asthma Symptoms, no Awakenings, and no As-needed Use)
Description: An asthma-control day was defined as a a night and day with no asthma symptoms, no awakenings due to asthma symptoms, and no as-needed medication use. The mean value from the treatment period was presented here.
Time Frame: 52-week treatment period
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Mean (Standard Deviation); unit: percentage of asthma-control days
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1033 | 1026
percentage of asthma-control days | 41.7 (37.3) | 37.9 (36.6)

13. Secondary Outcome: Asthma Control Questionnaire (ACQ)
Description: The ACQ developed by Juniper and colleagues (Juniper et al 1999) was used without the FEV1 and Beta 2-agonist questions. The Asthma Control Questionnaire has 5 questions that are assessed on a 7-point scale from 0 to 6 where 0 represents good control and 6 represents poor control. The overall score is the mean of the five responses. At least 4 out of the 5 questions must have been answered to provide a value. The mean of the overall score for Weeks 4 to 52 was presented here.
Time Frame: 4, 12, 24, 36 and 52 weeks after randomization
Population: The analysis set for efficacy was based on the full analysis set (FAS) in line with the ICH E9 guideline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Number analyzed (Participants) | 1040 | 1038
units on a scale | 1.162 (0.78) | 1.289 (0.75)

ADVERSE EVENTS:
Arm/Group | Symbicort SMART | Symbicort+Terbutaline As Needed
Serious Adverse Events (participants affected / at risk) | 41/1049 | 74/1042
Other Adverse Events (participants affected / at risk) | 279/1049 | 293/1042
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort SMART (N=1049) | Symbicort+Terbutaline As Needed (N=1042)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Cleft Lip (Congenital, familial and genetic disorders) | 1 | 0
Meniere's Disease (Ear and labyrinth disorders) | 1 | 0
Basedow's Disease (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Retinal Detachment (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Acute Abdomen (Gastrointestinal disorders) | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 1
Colonic Polyp (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric Polyps (Gastrointestinal disorders) | 0 | 1
Hernia Obstructive (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 2
Gastroenteritis (Infections and infestations) | 1 | 3
Tracheobronchitis (Infections and infestations) | 2 | 0
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 2 | 0
Acute Sinusitis (Infections and infestations) | 1 | 0
Breast Abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
H1n1 Influenza (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis Media Chronic (Infections and infestations) | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Tooth Abscess (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 | 2
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1
Sternal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast Cancer In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Abortion Threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature Baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Major Depression (Psychiatric disorders) | 1 | 0
Breast Calcifications (Reproductive system and breast disorders) | 0 | 1
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Infertility Male (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 31
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort SMART (N=1049) | Symbicort+Terbutaline As Needed (N=1042)
Nasopharyngitis (Infections and infestations) | 137 | 133
Bronchitis (Infections and infestations) | 69 | 77
Viral Upper Respiratory Tract Infection (Infections and infestations) | 60 | 72
Pharyngitis (Infections and infestations) | 49 | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other